CLINICAL TRIAL: NCT05621031
Title: Effects of Whole Body Vibration in Parkinson's Disease Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Seville (Other)
Collaborators: Asociación de Enfermos de Parkinson de Sevilla (Unknown)
Responsible Party: Principal Investigator, Paula González García, Principal investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USFISIOTERAPIAPGG01
Record Dates: First submitted 2022-11-03; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: parkinson disease,; whole body vibration; rigidity
MeSH Terms: conditions — Parkinson Disease; Muscle Rigidity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PDExperimental (Experimental): This group will receive usual care (physical therapy) and whole body vibration sessions.
  Interventions: Device: Whole body Vibration; Other: Habitual Therapy
- PDControl (Active Comparator): This group will receive usual care (physical therapy) and placebo whole body vibration session.
  Interventions: Other: Habitual Therapy; Device: Placebo whole body vibration

INTERVENTIONS:
Device: Whole body Vibration — Whole body vibration will be administered with a vibration platform (Power Plate Move). Subjects will do several exercises (squats and steps) whilst on the platform, set at these parameters: frequency 30 Hz; amplitude: 2 mm; 1 min activation; 1 min rest, 5 activations. 15 sessions will be carried out (2/week).
  Arms: PDExperimental
Other: Habitual Therapy — Physical therapy will be administered to all study subjects. Experimental group will perform their session the same day that the experimental intervention.
Device: Placebo whole body vibration — Placebo whole body vibration will be administered with a vibration platform (Power Plate Move). Subjects will do several exercises (squats and steps) whilst on the platform. The platform will only be working for 3 seconds (parameters: frequency 30 Hz; amplitude: 2 mm) and after 3 seconds, the vibration will stop. Same as experimental group, there will be 1 min placebo activation; 1 min rest, 5 activations. 15 sessions will be carried out (2/week).
  Arms: PDControl

SUMMARY:
The goal of this clinical trial is to know the effects of an intervention in Parkinson's disease symptoms. The main question it aims to answer are:

* Is whole body vibration able to reduce rigidity in Parkinson's participants?
* Can whole body vibration modify gait abilities and other Parkinson's symptoms? Participants (subjects with Parkinson's disease) will do habitual therapy treatment. Experimental group will also carry out whole body vibration sessions and control group will do placebo whole body vibration sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson Disease, in phase I and II according to Hoehn & Yahr phases.
* Able to maintain independently standing position.
* Able to understand instructions and score >24 in Minimental Test.

Exclusion Criteria:

* Changes in pharmacological treatment for PD symptoms during the study.
* Recent injuries in the last 12 weeks in lower limbs or trunk.
* Other neurological conditions not related to Parkinsonism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline muscle tone at 9 weeks | Week 9
  Muscle tone will be measured using Myoton Pro (Hz) in the following sites: plantar fascia, Achilles tendon, soleus, gastrocnemius, erector spinae (L3-L4, T12-L1, T8-T9,T3-T4 and C7-T1) , transversus abdominus, rectus femoris, infrapatellar tendon and anterior tibialis . Measures will be taken twice bilaterally.
Change from baseline muscle stiffness at 9 weeks | Week 9
  Muscle stiffness will be measured using Myoton Pro (N/m) in the following sites: plantar fascia, Achilles tendon, soleus, gastrocnemius, erector spinae (L3-L4, T12-L1, T8-T9,T3-T4 and C7-T1) , transversus abdominus, rectus femoris, infrapatellar tendon and anterior tibialis . Measures will be taken twice bilaterally.
Change from baseline muscle elasticity at 9 weeks | Week 9
  Muscle elasticity will be measured using Myoton Pro (logarithmic decrement) in the following sites: plantar fascia, Achilles tendon, soleus, gastrocnemius, erector spinae (L3-L4, T12-L1, T8-T9,T3-T4 and C7-T1) , transversus abdominus, rectus femoris, infrapatellar tendon and anterior tibialis . Measures will be taken twice bilaterally.
Change from week 9 muscle tone at 22 weeks (follow up period) | Week 22
  Muscle tone will be measured using Myoton Pro (Hz) in the following sites: plantar fascia, Achilles tendon, soleus, gastrocnemius, erector spinae (L3-L4, T12-L1, T8-T9,T3-T4 and C7-T1) , transversus abdominus, rectus femoris, infrapatellar tendon and anterior tibialis . Measures will be taken twice bilaterally.
Change from week 9 muscle stiffness at 22 weeks (follow up period) | Week 22
  Muscle stiffness will be measured using Myoton Pro (N/m) in the following sites: plantar fascia, Achilles tendon, soleus, gastrocnemius, erector spinae (L3-L4, T12-L1, T8-T9,T3-T4 and C7-T1) , transversus abdominus, rectus femoris, infrapatellar tendon and anterior tibialis . Measures will be taken twice bilaterally.
Change from week 9 muscle elasticity at 22 weeks (follow up period) | Week 22
  Muscle elasticity will be measured using Myoton Pro (logarithmic decrement) in the following sites: plantar fascia, Achilles tendon, soleus, gastrocnemius, erector spinae (L3-L4, T12-L1, T8-T9,T3-T4 and C7-T1) , transversus abdominus, rectus femoris, infrapatellar tendon and anterior tibialis . Measures will be taken twice bilaterally.
Changes from baseline gait functionality at 9 weeks | Week 9
  This outcome will be measured with the Modified Emory Functional Ambulation Profile. This scale assesses functional ambulation in terms of assistance and time under five different environmental conditions. Since time (seconds) if the main measure, there is not top score and the higher the score, the worse is the performance.
Changes from week 9 gait functionality at 22 weeks (follow up period) | Week 22
  This outcome will be measured with the Modified Emory Functional Ambulation Profile. This scale assesses functional ambulation in terms of assistance and time under five different environmental conditions. Since time (seconds) if the main measure, there is not top score and the higher the score, the worse is the performance.

SECONDARY OUTCOMES:
Changes from baseline thoracic kyphosis at 9 weeks | Week 9
  The degree of thoracic kyphosis will be measure with the mobile application Goniometer Pro (degrees). The mobile will the placed at T1 and T12 and will measure the angle between them.
Changes from week 9 thoracic kyphosis at 22 weeks (follow up period) | Week 22
  The degree of thoracic kyphosis will be measure with the mobile application Goniometer Pro (degrees). The mobile will the placed at T1 and T12 and will measure the angle between them.
Changes from baseline aspects of quality of life at 9 weeks | Week 9
  This outcome will be measured with the Parkinson's Disease Questionnaire (PDQ-399). This questionnaire assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living. The scores ranges between 0 and 800, with a lower score reflecting better quality of life.
Changes from week 9 aspects of quality of life at 22 weeks (follow up period) | Week 22
  This outcome will be measured with the Parkinson's Disease Questionnaire (PDQ-399). This questionnaire assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living. The scores ranges between 0 and 800, with a lower score reflecting better quality of life.
Changes from baseline freezing of gait at 9 weeks | Week 9
  This outcome will be measured with the Freezing of Gait Questionary. This scale assesses the severity and the frequency of the episodes of freezing during gait. It also considers the relationship of these episodes with other gait and motor aspects.The scores ranges between 0 and 24, with a lower score less freezing episodes.
Changes from week 9 freezing of gait at 22 weeks (follow up period) | Week 22
  This outcome will be measured with the Freezing of Gait Questionary. This scale assesses the severity and the frequency of the episodes of freezing during gait. It also considers the relationship of these episodes with other gait and motor aspects.The scores ranges between 0 and 24, with a lower score less freezing episodes.
Changes from baseline reactive balance at 9 weeks | Week 9
  This outcome will be measure with the section of reactive balance assessment of the Balance Evaluation System Test (BESTest). This section includes 5 items that specifically measures reactive balance and compensatory responses in all directions. The scores ranges between 0 and 18, with a lower score reflecting worse reactive balance.
Changes from week 9 reactive balance at 22 weeks | Week 22
  This outcome will be measure with the section of reactive balance assessment of the Balance Evaluation System Test (BESTest). This section includes 5 items that specifically measures reactive balance and compensatory responses in all directions. The scores ranges between 0 and 18, with a lower score reflecting worse reactive balance.

OTHER OUTCOMES:
Age | Baseline
  Years
Height | Baseline
  Cm
Weight | Baseline
  Kg
Time since Parkinson disease diagnosis | Baseline
  Years and months

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación de Enfermos de Parkinson de Sevilla, Seville, Spain